CLINICAL TRIAL: NCT02371850
Title: Determination of Plasma Nicotine Levels After Using Reference and Generic Transdermal Nicotine Patches With and Without Standardized Heat Application in Adult Smokers
Brief Title: Transdermal Patch CVD 1000: The Effect of Heat on Nicotine Release From Nicotine Patches in Adult Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Audra Stinchcomb, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00059146
Record Dates: First submitted 2015-02-06; First posted 2015-02-26 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Smoking
Keywords: Bioequivalence; Therapeutic Equivalency
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Intervention Model Description: Each subjects gets two procedure days with heating applied for one hour at hours 4 and hour 8 after the application of the Nicoderm CQ nicotine patch, then followed by two procedure days with heating applied for one hour at hours 4 and hour 8, after the application of the Aveva nicotine patch (total of four Procedure days)
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nicoderm patch first, then Aveva patch (Experimental): Each subject gets two procedure days with heating applied for one hour at hours 4 and hour 8 after the application of the Nicoderm CQ nicotine patch, then followed by two procedure days with heating applied for one hour at hours 4 and hour 8, after the application of the Aveva nicotine patch (total of four Procedure days)
  Interventions: Drug: Nicoderm patch first, then Aveva patch

INTERVENTIONS:
Drug: Nicoderm patch first, then Aveva patch — This is a single group assignment where each of 10 adult smokers completes 4 procedure days using a Nicoderm CQ nicotine patch (2 days) followed by the application of a generic Aveva patch (2 days). For each patch, heating is applied for one hour at hour 4 on the first procedure day and at hour 8 in the second procedure day (2 days per patch, or a total of 4 days per subject).
  Other Names: Brand name nicotine patch first, then generic nicotine patch

SUMMARY:
This is a single-dose, Open-label, Non-Randomized, 2-way Crossover Bioequivalence Study to compare nicotine release after heating of a brand name (Nicoderm CQ) and generic (Aveva skin patch) nicotine skin patches in adult smokers.

DETAILED DESCRIPTION:
This research study is intended to determine the effect of heat on FDA-approved nicotine transdermal patches and whether the heat applied will result in more nicotine being absorbed through the skin than without applying heat. This is important given that little is known about how the release of nicotine is affected by heat, particularly for generic products that are also available over the counter. This study will use nicotine patches (brand name and generic patches) that have been approved by the Food and Drug Administration (FDA) and are already sold over the counter to customers in the United States, and will not include any placebos.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men or non-pregnant women of any ethnic background between the age of 18 and 45 years old
* 2. Subjects should be cigarette smokers who smoke at least 5 cigarettes per day for one year or more.
* 3. Provide written informed consent before initiation of any study procedures.
* 4. Available for follow-up for the planned duration of the study
* 5. Able to communicate well with the investigators
* 6. Able to adhere to the study restrictions and examination schedule.
* 7. Subjects who are within their ideal body weight (BMI >17 and <= 25)
* 8. Demonstrate comprehension of the protocol procedures and knowledge of study by passing (>70% correct responses) a written examination containing 20 multiple choice and true false questions covering all aspects of the study including the purpose, procedures, risks and benefits.
* 9. Subjects deemed to be eligible as judged by the Medically Accountable Investigator (MAI) and determined by medical history, physical examination, and medication history.
* 10. Have a normal blood pressure (systolic: 90-140 mmHg; diastolic: 50-90 mmHg) and heart rate (55-100 bpm),
* 11. Have normal screening laboratories for WBC, Hgb, platelets, sodium, potassium, chloride, bicarbonate, BUN, creatinine, ALT and AST
* 12. Have normal screening laboratories for urine protein and urine glucose.
* 13. Female subjects must be of non-childbearing potential (as defined as surgically sterile [i.e. history of hysterectomy or tubal ligation] or postmenopausal for more than 1 year), or if of childbearing potential, must be non-pregnant at the time of enrollment and on the morning of each procedure day, and must agree to use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner.
* 14. Agrees not to participate in another clinical study during the study period.
* 15. Agrees not to donate blood to a blood bank throughout participation in the study and for at least 3 months after last procedure day.
* 16. Have a normal ECG
* 17. Be a smoker willing to refrain from smoking 10 hours prior to, and during, each procedure day of the study.

Exclusion Criteria:

* 1. Subjects who are nonsmokers or smoke less than 5 cigarettes per day
* 2. Women who are pregnant or lactating or have a positive serum pregnancy test at enrollment or on the morning of any procedure day.
* 3. Participation in any ongoing investigational drug trial or clinical drug trial
* 4. Abnormal Vital signs, defined as:

  * Hypertension (systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg) at rest on 2 separate days)
  * Heart rate <55 at rest on 2 separate days
  * Respiratory rate >20
* 5. Temperature > 38.0 ºC (100.4 ºF) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 7 days of administration of the transdermal patch.
* 6. Active positive Hepatitis B, C, and HIV serologies
* 7. Positive urine drug screening test
* 8. Use of any prescription medication during the period 0 to 30 days or over-the counter medication (vitamin, herbal supplements and birth control medications not included) during the period 0 to 5 days before entry to the study
* 9. Donation or loss of greater than one pint of blood within 60 days of entry to the study
* 10. Any prior serious adverse reaction or hypersensitivity to nicotine or any of the inactive ingredients in the patch (acrylate adhesive, polyester, silicone, ethylene vinyl acetate-copolymer polyisobutylene and polyethylene)
* 11. Have a diagnosis of schizophrenia or other major psychiatric diagnosis.
* 12. Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month before enrollment in this study or expects to receive an experimental agent during the study.
* 13. Any condition that would, in the opinion of the Medically Accountable Investigator (MAI), place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* 14. Inability to communicate or co-operate with the investigators
* 15. History of consumption of alcohol within 24 hours prior to dose administration
* 16. Scarring on upper arms, including tattoos at planned site of patch placement making skin reactions not evaluable
* 17. Subject who currently has any of the following conditions:

  1. Thrombophlebitis, thromboembolic disorders
  2. A past history of deep vein thrombophlebitis or thromboembolic disorders
  3. Cerebrovascular or coronary artery disease (current or past history)
  4. Valvular heart disease with complications
  5. Severe hypertension
  6. Diabetes with vascular involvement
  7. Headaches with focal neurological symptoms
  8. Major surgery with prolonged immobilization
* 18. Medical history of a serious chronic condition (e.g. allergic conditions such as anaphylaxis, asthma or generalized drug reaction).
* 19. Medical history of significant dermatologic diseases or conditions, such as atopy, psoriasis, vitiligo or conditions known to alter skin appearance or physiologic response (e.g. diabetes, porphyria).
* 20. History of significant dermatologic cancers (e.g. melanoma, squamous cell carcinoma), except basal cell carcinomas that were superficial and did not involve the investigative site.
* 21. Within 10 hours prior to dosing, use of other nicotine products (e.g. nicotine gum or other nicotine-containing products) that would significantly influence or exaggerate responses to the nicotine patches used in this study.
* 22. Within 72 hours prior to dosing, use of antihistamines or use of topical drugs at patch site.
* 23. Subject has an obvious difference in skin color between arms or the presence of a skin condition, open sores, scar tissue, tattoo, or coloration that would interfere with placement of test articles, skin assessment, or reactions to drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samer El-Kamary, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore Center for Vaccine Development, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicoderm Patch First, Then Aveva Patch: Each subjects gets two procedure days with heating applied for one hour at hours 4 and hour 8 after the application of the Nicoderm CQ nicotine patch, then followed by two procedure days with heating applied for one hour at hours 4 and hour 8, after the application of the Aveva nicotine patch (total of four Procedure days)
Period: Overall Study
Arm/Group | Nicoderm Patch First, Then Aveva Patch
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nicoderm Patch First, Then Aveva Patch
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Maximum Serum Concentration (Cmax)
Description: The main outcome measure of the study is the measurement of maximum serum concentration (Cmax)
Time Frame: four procedure days for each participant
Population: Ten adult smokers between 24 and 44 years of age at the time of enrollment completed the study. The clinical study was an single-group, open-label study. Each subject completed 4 study visits where in-vivo nicotine levels were measured using a reference patch (Nicoderm CQ) and a generic patch (Aveva)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nicoderm Patch First, Then Aveva Patch
Number analyzed (Participants) | 10
ng/mL
  NicoDerm CQ early heat serum nicotine Cmax | 27.47 (10.49)
  Aveva early heat serum nicotine Cmax | 21.32 (13.42)
  NicoDerm CQ late heat serum nicotine Cmax | 28.04 (8.98)
  Aveva late heat serum nicotine Cmax | 22.96 (9.55)

2. Secondary Outcome: AUC
Description: (area under the concentration-time curve of nicotine 0-12 h)
Time Frame: 0-12 h for each of the four procedure day
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- NicoDerm CQ (Early Heat); Aveva (Early Heat): early heat
- NicoDerm CQ (Late Heat); Aveva (Late Heat): late heat
Arm/Group | NicoDerm CQ (Early Heat) | NicoDerm CQ (Late Heat) | Aveva (Early Heat) | Aveva (Late Heat)
Number analyzed (Participants) | 10 | 10 | 10 | 10
h*ng/mL | 173.8 (54.10) | 184.3 (67.92) | 116.3 (73.41) | 121.20 (49.98)

ADVERSE EVENTS:
Time Frame: 1 year
Description: The definition does not differ.
Groups:
- Nicoderm Patch 4 h Heat Application; Nicoderm Patch 8 h Heat Application; Aveva Patch 4 h Heat Application; Aveva Patch 8 h Heat Application: Each subjects gets two procedure days with heating applied for one hour at hours 4 and hour 8 after the application of the Nicoderm CQ nicotine patch, then followed by two procedure days with heating applied for one hour at hours 4 and hour 8, after the application of the Aveva nicotine patch (total of four Procedure days)
Arm/Group | Nicoderm Patch 4 h Heat Application | Nicoderm Patch 8 h Heat Application | Aveva Patch 4 h Heat Application | Aveva Patch 8 h Heat Application
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 6/10 | 7/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicoderm Patch 4 h Heat Application (N=10) | Nicoderm Patch 8 h Heat Application (N=10) | Aveva Patch 4 h Heat Application (N=10) | Aveva Patch 8 h Heat Application (N=10)
Erythema at the site of patch placement (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Elevated Respiratory Rate (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 4 (5) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — at IV site
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — pruritus at patch application site
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heat rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — due to heating pad application
Numbness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — (transient) right thumb
Skin redness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — TDS site (due to external heat application)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Elevated systolic (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restricted until the manuscript is published in a peer-reviewed journal.